CLINICAL TRIAL: NCT01046227
Title: Antibody Titer Analysis Afer Monovalent Vaccination in Pediatric Haemato-oncology Patients
Brief Title: Antibody Titer Analysis After H1N1 Vaccination in Pediatric Haemato-oncology Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 200912031R
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2009-12

CONDITIONS: Serology Analysis; Novel H1N1 Influenza Vaccination; Pediatric Haemato-oncology Patients
Keywords: Serology; Monovalent inactivated H1N1 vaccine; Pediatric haemato-oncology patients
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum for serology of H1N1 antibody Nasopharyngeal or oropharyngeal swab for Novel H1N1 PCR
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Serology after Novel H1N1 vaccination: This study is designed to investigate the antibodies titers before and after the novel H1N1 influenza vaccination in pediatric haemato-oncology patients.
  Interventions: Biological: Influenza A (H1N1) 2009 monovalent vaccine, inactivated

INTERVENTIONS:
Biological: Influenza A (H1N1) 2009 monovalent vaccine, inactivated — Serology study before and after Influenza A (2009) monovalent vaccine, inactivated
  Other Names: Influenza Virus Vaccine, AdimFlu-S (A/H1N1)

SUMMARY:
The patients of pediatric haemato-oncology have a higher risk for novel H1N1 influenza infection than general population, and they are strongly recommended to receive novel H1N1 vaccination. However, there is no previous data to answer how the efficacy and effectiveness of novel H1N1 vaccination is in patients of pediatric haemato-oncology. This study is designed to investigate the antibodies titers before and after the novel H1N1 influenza vaccination in these patients. Titer of H1N1 influenza virus antibodies will be determined by hemagglutinin inhibition assay (HAI). A HAI titer with a 4-fold rise or greater is defined as seroconversion. Study subjects with seroconversion are regarded as responsiveness to the vaccination. Meanwhile, if the patient presents influenza-like symptoms, we will perform throat swab or nasal swab for influenza rapid test, viral isolation, and novel H1N1 influenza PCR to confirm the diagnosis. After the study, we will be able to know whether or not current novel H1N1 influenza vaccination schedule is adequate and efficient for pediatric haemato-oncology patients.

DETAILED DESCRIPTION:
The emergence of novel H1N1 influenza in 2009 has a great impact to the societies in Taiwan and worldwide. The patients of pediatric haemato-oncology have a higher risk for novel H1N1 influenza infection than general population, and they are strongly recommended to receive novel H1N1 vaccination. However, there is no previous data to answer how the efficacy and effectiveness of novel H1N1 vaccination is in patients of pediatric haemato-oncology. This study is designed to investigate the antibodies titers before and after the novel H1N1 influenza vaccination in these patients. Thus two blood samples will be drawn. The first sample will be collected before the vaccination and the second one will be collected three weeks after the vaccination (If the patient is younger than 9 years old, the third sample will be collected three weeks after the booster vaccination). Titer of H1N1 influenza virus antibodies will be determined by hemagglutinin inhibition assay (HAI). A HAI titer with a 4-fold rise or greater is defined as seroconversion. Study subjects with seroconversion are regarded as responsiveness to the vaccination. We will analyze seroconversion rate as well. Meanwhile, if the patient presents influenza-like symptoms, we will perform throat swab or nasal swab for influenza rapid test, viral isolation, and novel H1N1 influenza PCR to confirm the diagnosis. After the study, we will be able to know whether or not current novel H1N1 influenza vaccination schedule is adequate and efficient for pediatric haemato-oncology patients.

ELIGIBILITY:
Inclusion Criteria:

* Boys or girls aged ≧ 6 months old to 18 years old on the day of first vaccination;
* Subject and/or parents(s)/legal guardian(s) was willing to comply with planned study procedures and be available for all study visits;
* Subject was ever treated at pediatric haemato-oncology ward
* Subject and/or parents(s)/legal guardian(s) must read and signed the study-specific informed consent prior to initiation of any study procedure.

Exclusion Criteria:

* History of hypersensitivity to eggs or egg protein or similar pharmacological effects to study medication (AdimFlu-S (A/H1N1));
* Personal or family history of Guillain-Barré Syndrome;
* An acute febrile illness within the last 72 hours prior to vaccination;
* Subject with bleeding disorder or has any coagulation disorder that needs receipt of anticoagulants in the 3 weeks preceding inclusion contraindicating intramuscular injection;
* Subjects with influenza-like illness as defined by the presence of fever (temperature ≧38.5℃ ) and at least two of the following four symptoms: headache, muscle/joint aches and pains (e.g. myalgia/arthralgia), sore throat and cough;
* Female subjects who are pregnant, lactating or likely to become pregnant during the study; Women of childbearing potential disagree to use an acceptable method of contraception (e.g., hormonal contraceptives, IUD, barrier device or abstinence) throughout the study;
* Underlying condition in the investigator's opinion may be inappropriate for vaccination;

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study is designed to investigate the antibodies titers before and after the novel H1N1 influenza vaccination in pediatric haemato-oncology patients.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-02 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
This study is designed to investigate the antibodies titers before and after the novel H1N1 influenza vaccination in these patients. Titer of H1N1 influenza virus antibodies will be determined by hemagglutinin inhibition assay (HAI). | Dec, 2009 - Feb, 2010

SECONDARY OUTCOMES:
If the patient presents influenza-like symptoms during the six month follow up period, we will perform throat swab or nasal swab for influenza rapid test, viral isolation, and novel H1N1 influenza PCR to confirm the diagnosis. | Dec, 2009 - Jun, 2010

CONTACTS AND LOCATIONS:
Overall Officials: Luan-Yin Chang, MD, Principal Investigator — National Taiwan University Hospital, Taipei, Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan